CLINICAL TRIAL: NCT06796231
Title: Evaluation of the Efficacy and Prognosis of PD-1 Monoclonal Antibody in the Treatment of the Skin and Subcutaneous Tissue Phaeohyphomycosis of Immunodeficient Patients
Brief Title: Efficacy of PD-1 Monoclonal Antibody in the Treatment of Phaeohyphomycosis
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Lu Sha, Principal Investigator（Lu Sha）, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-823-01
Record Dates: First submitted 2024-11-16; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Phaeohyphomycosis
MeSH Terms: conditions — Phaeohyphomycosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Phialophora verrucosa
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective was to evaluate the clinical efficacy of PD-1 inhibitor (PD-1 monoclonal antibody) in the treatment of skin and subcutaneous mucocytosis infection, including the comparison of immune cell groups before and after treatment, the changes in the proportion of CD4+T cells and CD8+T cells, and the changes in the inflammatory cytokines of the serum after co-culture of human peripheral blood mononuclear cells (PBMC) with fungi before and after treatment. The improvement of lesions and the relief of symptoms. The secondary objective is to evaluate the safety of PD-1 inhibitors during treatment, including monitoring and recording all adverse events and immune-related adverse reactions.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the clinical efficacy of PD-1 inhibitors (PD-1 monoclonal antibodies) in the treatment of skin and subcutaneous mucocytosis infections. This included comparing immune cell groups before and after treatment, observing changes in the proportion of CD4+ T cells and CD8+ T cells, and monitoring alterations in serum inflammatory cytokines following co-culture of human peripheral blood mononuclear cells (PBMCs) with fungi before and after treatment. Additionally, the study assessed the improvement of lesions and the relief of symptoms. The secondary objective was to evaluate the safety of PD-1 inhibitors during treatment, which involved monitoring and recording all adverse events and immune-related adverse reactions.

The study confirmed that the expression of co-inhibitory molecules is upregulated in exhausted T cells following chronic infection. Blocking the expression of these co-inhibitory molecules may be significant in the treatment of such diseases, providing potential theoretical support for understanding the underlying mechanisms and developing subsequent new therapeutic approaches.

Integrating the above information, we can conclude the following:

1. Clinical Efficacy Assessment: By comparing immune cell groups, T cell subsets, and serum inflammatory cytokines before and after treatment with PD-1 inhibitors, the study aimed to evaluate the effectiveness of PD-1 inhibitors in the treatment of skin and subcutaneous infections, as well as observing improvements in lesions and symptom relief.
2. Safety Assessment: Monitoring and recording all adverse events and immune-related adverse reactions during the treatment period to assess the safety of PD-1 inhibitors.
3. Immune Mechanism Exploration: The study found that the expression of co-inhibitory molecules is upregulated in exhausted T cells following chronic infection, indicating that blocking the expression of these molecules may play a positive role in treating such diseases, offering a new perspective for future treatment strategies.
4. Theoretical Support: The results of this study provide a theoretical basis for understanding the immune mechanisms of chronic infections and potential support for developing new therapeutic approaches, which is significant for improving patient outcomes and developing new therapies.

In summary, the study not only assessed the efficacy and safety of PD-1 inhibitors but also provided valuable information for深入 understanding the immune mechanisms of chronic infections and developing new treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* A. Fungal infection of skin and subcutaneous tissue; b, the conventional treatment effect is not good; c, immunodeficient host; d. PD-1 has been used or is intended to be used for treatment

Exclusion Criteria:

* Severe autoimmune disease; b, serious heart and lung disease, liver and kidney insufficiency; c. Lactating women and pregnant women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Fungal infection of skin and subcutaneous tissue;
  2. the conventional treatment effect is not good;
  3. immunodeficient host; d. PD-1 has been used or is intended to be used for treatment
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-07-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Changes in CD4 T cells and CD8 T cells | through study completion, an average of 1 month
  Changes in CD4 T cells and CD8 T cells：through study completion, an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangdong, GuangZhou, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR